CLINICAL TRIAL: NCT07197645
Title: A Phase 1 Pharmacokinetic, Dosimetry, Safety, and Dose Optimization Study for a Single Dose of TLX090-Tx (153SmDOTMP) to Treat Metastatic Bone Pain
Brief Title: Samarium Optimized for Long-lasting Analgesia in Cancerous End-stage Bone Pain
Acronym: SOLACE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 153Sm-TLX090-101
Record Dates: First submitted 2025-07-30; First posted 2025-09-29 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Bone Pain; Metastatic Bone Tumor; Bone Metastases in Subjects With Advanced Cancer
Keywords: samarium; radioligand; radioisotope; metastatic bone pain palliation; Samarium-153; DOTMP; bone-seeking radiopharmaceutical
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part A - Cohort 1 (Experimental): Dose Escalation
  Interventions: Drug: 153Sm-DOTMP

INTERVENTIONS:
Drug: 153Sm-DOTMP — TLX090-Tx will be administered as a single ascending intravenous dose to participants with at least 1 confirmed painful osteoblastic bone tumor that exhibits avid uptake as shown by 99mTcdiphosphonate bone scans undertaken within 60 days of dosing.

SUMMARY:
This is an open label, 2-part early phase study designed to evaluate the safety, pharmacokinetics, radiation dosimetry, and preliminary efficacy of TLX090-Tx in patients with painful bone metastases.

ELIGIBILITY:
Inclusion Criteria:

* Participants have had disease progression while on anti-cancer treatment, and are not eligible for the treatments, or their lesions are not amenable to palliative EBRT.
* Participants must have a histologically confirmed diagnosis of malignancy at any time prior to their participation in this clinical trial with multiple metastatic bone lesions with at least 1 metastatic painful osteoblastic tumor that causes a minimum pain score of 4 on the NRS11.
* Participants must have bone cancer in one or more skeletal locations as identified by a 99mTc-diphosphonate bone scan within 60 days of dosing. At least one lesion must be osteoblastic. If described as osteosclerotic, radiology confirmation that the lesion is osteoblastic is required. Adequate organ function, including:
* Renal function, defined as a measured creatinine clearance (CrCl) ≥30 mL/min as per Cockroft Gault or based on radioisotope glomerular filtration rate (GFR).
* Hematologic function, defined as a platelet count of >100,000 cells/mm3 and an Absolute neutrophil count (ANC) of >1000 cells/mm3.
* Hemoglobin ≥8 g/dL.
* Liver function:
* Total bilirubin ≤1.5 × the upper limit of normal (ULN).
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤5 × ULN with participants with known liver metastases.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤3 × ULN with participants with Gilbert's Syndrome.
* Life expectancy of at least 16 weeks from the date of study drug administration (Day 1).
* Karnofsky performance status >60%, assessed during the screening period prior to study drug administration.

Exclusion Criteria:

* Participants are pregnant or breastfeeding.
* Participants who have received maximum tolerable radiation to the spinal cord, have untreated pathologic bone fracture, spinal cord compression, unstable spine, or imminent long bone fracture.
* Participants with a bone scan pattern showing diffuse, intense skeletal uptake with absent or faint kidney / bladder activity, typically indicating widespread bone metastases or high bone turnover from metabolic or hematologic diseases (Superscan) pattern on Technetium 99-m bone scan scintigraphy - defined as diffusely increased skeletal uptake with absent or markedly reduced renal and soft tissue visualization - are excluded from the study.
* Participants with impending or suspected or at high risk for spinal cord compression.
* Participants with neurogenic pain or significant pain associated with soft tissue lesions or other pain that, in the opinion of the Investigator, might interfere with the assessment of pain relief for bone tumors.
* Participants who require surgery over their trial period that would require pain medication or analgesia.
* Clinically significant illness or clinically relevant trauma within 2 weeks before the administration of the investigational product.
* History of unstable angina (defined as angina at rest) or new-onset angina diagnosed within the 3 months prior to screening.
* History of myocardial infarction within 3 months prior to screening, as determined by medical history / Baseline ECG.
* Uncontrolled cardiac arrhythmias (≥Grade 3 CTCAE version 5.0) or any history of ≥Grade 3 arrhythmia.
* Congestive heart failure ≥New York Heart Association Class 2.
* Clinically significant abnormalities on ECG at screening including corrected QT interval (Fridericia's formula) >450 msec for males or 470 msec for females at screening.
* Inability to complete the needed investigational and standard imaging examinations due to any reason (eg, severe claustrophobia, inability to lie still for the entire imaging time).
* Presence of any other condition that may increase the risk associated with study participation or interfere with the interpretation of study results, and, in the opinion of the study Investigator, would make the participant inappropriate for entry into the study.
* Participants with active infections (human immunodeficiency virus, human papillomavirus. Hepatitis A, Hepatitis B, and Hepatitis C).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2027-04-26 (Estimated); Study Completion 2027-07-05 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) [Safety and Tolerability] | Up to 6 weeks post-dose
  Incidence and severity of hematologic and non-hematologic toxicities, graded per CTCAE v5.0, assessed through 6 weeks post-dose.

SECONDARY OUTCOMES:
Change from baseline in patient-reported bone pain severity using the NRS-11 scale on the form | Baseline to 16 weeks post-dose
  Change in pain score using NRS-11, assessed up to 16 weeks post-dose.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Houston Metro Urology, Houston, Texas
  - Oncology Consultants, Houston, Texas
  - Excel Diagnostics and Nuclear Oncology Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No